CLINICAL TRIAL: NCT06323265
Title: A Real-world Study of Adebrelimab Combined With Chemotherapy±Chest Radiotherapy in Patients With Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, Study Principal Investigator, Hebei Medical University Fourth Hospital
Other Study IDs: ARL-SCLC-001
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental
  Interventions: Drug: Adebrelimab + chemotherapy; Radiation: ±chest radiotherapy

INTERVENTIONS:
Drug: Adebrelimab + chemotherapy — Adebrelimab: 1200mg, d1, iv (30-60min), Q3W ,up to progressive disease or toxicity intolerable Chemotherapy: etoposide 100mg/m2，d1-3，iv；carboplatin AUC=5-6，d1，iv；or cisplatin 75mg/m2，d1，iv，Q3W，4 cycles；
Radiation: ±chest radiotherapy — Chest radiotherapy: 3Gy/15f-18f or 2Gy/20f-25f

SUMMARY:
The purpose of this study is to assess efficacy and safety of patients who receive Adebrelimab combined with chemotherapy±chest radiotherapy as first-line treatment of extensive stage small cell lung cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age:≥18 years old;
2. Patients with extensive stage small cell lung cancer confirmed by histopathology;
3. Normal function of major organs;
4. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Patients with drug allergy sufferers;
2. Serious and uncontrolled organic lesions or infections, such as decompensated heart, lung, kidney failure, etc;
3. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
4. The researchers think inappropriate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: extensive stage small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured stable disease
Disease control rate (DCR) | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured progressive disease
Duration of Overall Response（DoR） | tumor assessment every 6 weeks since the treatment began，up to 24 months
  The duration of overall response is measured from the time that measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented
Overall survival (OS) | the first day of treatment to death or last survival confirm date,up to 24 months
  Baseline to measured date of death from any cause
Adverse events | up to 24 months
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. The number of Participants with adverse events will be recorded at each treatment visit

CONTACTS AND LOCATIONS:
Locations (1):
- Jun Wang, Shijiazhuang, Hebei, China